CLINICAL TRIAL: NCT01829854
Title: Unrecognised Obstructive Sleep Apnoea In Cardiac Surgery Patient In The Asian Population
Brief Title: To Investigate the Incidence of Obstructive Sleep Apnoea in Patient Undergoing Open Heart Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Other Study IDs: RG423-12HTM
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Obstructive Sleep Apnoea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a study to investigate the incidence of Obstructive Sleep Apnoea in Patient undergoing open heart Surgery . This will include enrolment of 400 patient undergoing open heart surgery .

ELIGIBILITY:
Inclusion Criteria:

* adults male and female , aged 45 years old and above
* undergoing open heart surgery that requires hospital stays of more than 5 days

Exclusion Criteria:

* previous diagnosis and treatment of OSA or any sleep related breathing disorder.
* unwilling or physically unavailable for polysomnography before surgery.
* Patient undergoing MAZE procedure .
* Patient with severe COPD

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient undergoing open heart surgery and is more than 45 years old . These patient are also required to stay in hospital for more than 5 days .
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-12 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Obstructive Sleep Apnoea | 2 years
  To look at the incidence of Obstructive Sleep Apnoea in Patient undergoing open heart Surgery .

CONTACTS AND LOCATIONS:
Overall Officials: Sivakumar Krishnasamy, MD, MMed(Surgery), Principal Investigator — University of Malaya
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia